CLINICAL TRIAL: NCT06850142
Title: A Comparative Study Between TMJ Discopexy to External Ear Cartilage Versus to Temporal Fascia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Collaborators: Sohag University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, Prof. Oral & Maxillofacial Surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMJ discopexy
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Joint Disc Displacement; Temporomandibular Joint Disc Displacement, Without Reduction
Keywords: External ear cartilage; Anterior disc displacement without reduction.; Temporal fascia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- discopexy of Temporo-mandibular joint (TMJ) disc to external ear cart (Experimental): 30 patients underwent discopexy of Temporo-mandibular joint (TMJ) disc to external ear cartilage
  Interventions: Procedure: Discopexy to external ear cartilage
- discopexy of TMJ disc to temporal fascia. (Active Comparator): Patients underwent discopexy of TMJ disc to temporal fascia.
  Interventions: Procedure: Discopexy to temporal fascia

INTERVENTIONS:
Procedure: Discopexy to external ear cartilage — stabilizing the articular disc within the temporomandibular joint (TMJ) in patients experiencing TMJ disorders (TMD) to external ear cartilage
  Arms: discopexy of Temporo-mandibular joint (TMJ) disc to external ear cart
Procedure: Discopexy to temporal fascia — stabilizing the articular disc within the temporomandibular joint (TMJ) in patients experiencing TMJ disorders (TMD) to temporal fascia
  Arms: discopexy of TMJ disc to temporal fascia.

SUMMARY:
Discopexy is a surgical procedure aimed at stabilizing the articular disc within the temporomandibular joint (TMJ) in patients experiencing TMJ disorders (TMD). The TMJ is a complex joint responsible for jaw movement, and its proper function relies on the alignment and stability of the articular disc, a fibrocartilaginous structure that cushions the joint. In cases of disc displacement or dysfunction, patients may experience pain, clicking, limited jaw movement, and other symptoms.

DETAILED DESCRIPTION:
Discopexy involves repositioning and securing the displaced disc to its anatomical position, often using sutures or anchors, to restore normal joint mechanics and alleviate symptoms. This procedure is typically considered when conservative treatments, such as physical therapy or splints, have failed to provide relief. Discopexy aims to improve joint function, reduce pain, and prevent further degenerative changes in the TMJ. The aim of the present study is to compare between new surgical techniques of discopexy of TMJ disc either to external ear cartilage or to temporal fascia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary TMD with complete anterior disc displacement without reduction with no or minimal osteoarthritic changes

Exclusion Criteria:

* osteoarthritis

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | baseline, 1 month, 3 months, 6 months
  The Visual Analog Scale (VAS) It consists of a straight line, typically 10 centimeters (100 mm) in length, with one end labeled "No Pain" and the other end labeled "Worst Pain Imaginable."

SECONDARY OUTCOMES:
Disc position | baseline, 1 month, 3 months, 6 months
  assess the position of the articular disc in the TMJ either Normal, anterior displacement (with or without reduction), posterior displacement, or lateral displacement.
Maximum Mouth opening | baseline, 1 month, 3 months, 6 months
  used to assess the functional capacity of the temporomandibular joint (TMJ) and the surrounding musculoskeletal structures.

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa shabaan, PhD, Principal Investigator — Fayoum University
Locations (1):
- Faculty of Dentistry- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez LV, Lopez JP, Orjuela MP, de la Sen O, Diaz-Baez D, Martin-Granizo R. Could temporomandibular joint arthroscopic discopexy with resorbable pins or disc mobilisation influence mandibular condyle marrow? Br J Oral Maxillofac Surg. 2025 Jan;63(1):39-46. doi: 10.1016/j.bjoms.2024.10.226. Epub 2024 Oct 10. PMID 39592295
- [Result] Jerez-Frederick D, Albers D, Fuenzalida C, Laissle G, Avila-Oliver C. Is the Complexity of Arthroscopic Temporomandibular Joint Surgery Associated With Short-Term Complication Rates? J Oral Maxillofac Surg. 2025 Mar;83(3):270-278. doi: 10.1016/j.joms.2024.11.008. Epub 2024 Nov 20. PMID 39645229
- [Result] Renapurkar SK. Discectomy Versus Disc Preservation for Internal Derangement of the Temporomandibular Joint. Oral Maxillofac Surg Clin North Am. 2018 Aug;30(3):329-333. doi: 10.1016/j.coms.2018.05.002. Epub 2018 Jun 7. PMID 29885876